CLINICAL TRIAL: NCT01170884
Title: Comparing Safety and Efficacy of Combigan® and Lumigan® With Lumigan® Alone in Glaucoma or Ocular Hypertension Subjects Treated With Xalatan®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-COM-09-013
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Results first posted 2012-01-12 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Timolol; Ophthalmic Solutions; Bimatoprost; Brimonidine Tartrate, Timolol Maleate Drug Combination; Hypromellose Derivatives

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Combigan® + Lumigan® (Active Comparator): COMBIGAN® (fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution) adjunctive to LUMIGAN® (bimatoprost 0.03% ophthalmic solution)
  Interventions: Drug: fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution; bimatoprost 0.03% ophthalmic solution
- Lumigan® (Active Comparator): LUMIGAN® (bimatoprost 0.03% ophthalmic solution) plus Gen Teal® Mild (hypromellose 0.2% eye drops) used for masking purposes
  Interventions: Drug: bimatoprost 0.03% ophthalmic solution; hypromellose 0.2% eyedrops

INTERVENTIONS:
Drug: fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution; bimatoprost 0.03% ophthalmic solution — 1 drop of fixed combination of brimonidine tartrate 0.2% timolol maleate 0.5% ophthalmic solution (Combigan®) taken approximately 12 hours apart, up to 2 times a day and 1 drop of bimatoprost 0.03% ophthalmic solution (Lumigan®) taken once every 24 hours.
  Other Names: COMBIGAN®; LUMIGAN®
  Arms: Combigan® + Lumigan®
Drug: bimatoprost 0.03% ophthalmic solution; hypromellose 0.2% eyedrops — 1 drop of bimatoprost 0.03% ophthalmic solution (Lumigan®) taken approximately every 24 hours; mild lubricant eyedrops (Gen Teal® Mild) for masking purposes
  Other Names: LUMIGAN®; Gen Teal® Mild
  Arms: Lumigan®

SUMMARY:
Comparing Safety and Efficacy of Combigan® and Lumigan® with Lumigan® Alone in Glaucoma or Ocular Hypertension Subjects Treated with Xalatan®.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with glaucoma or ocular hypertension.
* Visual Acuity 20/100 or better in both eyes

Exclusion Criteria:

* Any active ocular disease
* History of any intraocular surgery or glaucoma laser surgery within 3 months
* Contraindication to pupil dilation
* Use of topical, periorbital, intravitreal, or systemic steroid within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Dallas, Texas, United States

REFERENCES:
- [Background] Myers JS, Vold S, Zaman F, Williams JM, Hollander DA. Bimatoprost 0.01% or 0.03% in patients with glaucoma or ocular hypertension previously treated with latanoprost: two randomized 12-week trials. Clin Ophthalmol. 2014 Mar 27;8:643-52. doi: 10.2147/OPTH.S59197. eCollection 2014. PMID 24707169

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combigan® + Lumigan® | Lumigan®
Started | 59 | 62
Completed | 54 | 60
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combigan® + Lumigan® | Lumigan® | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.52) | 62.6 (13.19) | 63.3 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 64
  Male | 31 | 26 | 57

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal Intraocular Pressure (IOP) at Week 12
Description: Mean Diurnal (average of 8 AM, 10 AM, and 4 PM time points) IOP at Week 12 in the study eye. IOP is a measurement of the fluid pressure inside the eye.
Time Frame: Week 12
Population: Intent-to-Treat (ITT) included all subjects who were randomized to study medication.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mm Hg)
Arm/Group | Combigan® + Lumigan® | Lumigan®
Number analyzed (Participants) | 59 | 62
Millimeters of mercury (mm Hg) | 15.4 (2.34) | 19.2 (3.42)

ADVERSE EVENTS:
Arm/Group | Combigan® + Lumigan® | Lumigan®
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/62
Other Adverse Events (participants affected / at risk) | 10/59 | 1/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combigan® + Lumigan® (N=59) | Lumigan® (N=62)
Foreign Body Sensation (Eye disorders) | 3 | 0
Ocular Redness (Eye disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo